CLINICAL TRIAL: NCT07379099
Title: Implementation of the Personalized Care Plan (PCP) Proposed at the End of Step 2 of the ICOPE Program : Description of the Procedures for Negotiating the PCP With the Patient, the Procedures for Implementing the PCP in a Multi-professional Setting, and Implementation of the PCP at 1 Year
Brief Title: Implementation of the Personalized Care Plan (PCP) Proposed at the End of Step 2 of the ICOPE Program
Acronym: INEPPS
Status: Recruiting | Type: Observational
Sponsor: MSPU de Pins-Justaret (Other)
Responsible Party: Sponsor
Other Study IDs: INEPPS
Record Dates: First submitted 2026-01-23; First posted 2026-01-30 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Frailty; Frailty at Older Adults
MeSH Terms: conditions — Frailty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The ICOPE (Integrated Care for the Elderly) program is based on an integrated approach including a personalized care plan (PCP). Negotiation methods with the patient and interprofessional cooperation could be key elements in the success of this program. The main objective is to evaluate the feasibility of the implementation of the ICOPE program on the number and content of the PCP carried out at 1 year

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 60 years
* ADL ≥ 5.5
* Affiliated or beneficiary of a social security scheme or equivalent.
* having completed a STEP 2 ICOPE
* not opposed to the collection of their data

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Older adults aged 60 years and above, functionally independent
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2027-06-01 (Estimated); Study Completion 2028-04-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of PCP completed | At 12 months
  Proportion of personalized care plan (PCP) completed

CONTACTS AND LOCATIONS:
Locations (1):
- Maison de santé des Fontaines, Toulouse, France